CLINICAL TRIAL: NCT00780936
Title: Effect of Peripheral Nerve Block on Inflammatory and Nociceptive Biomarkers in a UV-B Burn Model in Humans
Brief Title: Effects of a Peripheral Nerve Block on Biomarkers of Pain and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SU-01222008-984; eProtocol number 10740
Record Dates: First submitted 2008-10-24; First posted 2008-10-28 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain

INTERVENTIONS:
Procedure: femoral nerve block

SUMMARY:
The purpose of this study is to determine the effect of a local anesthetic nerve block on markers of inflammation and pain after a sunburn. This is important because it may provide information regarding the way that nerve blocks help with the treatment of pain and in particular provide preemptive analgesia.

ELIGIBILITY:
Inclusion Criteria:1. Between 18 and 50 years of age 2. Fluent in English language 3. Provide written informed consent 4. Skin pigmentation type II or III
 Exclusion Criteria:1. Current use of prescription drugs interfering with study objective 2. Use of over-the-counter analgesic/anti-inflammatory drugs within 48h of study participation 3. Current acute or chronic pain conditions 4. Significant medical conditions including psychiatric, neurological, and dermatological diseases 5. Pregnancy 6. Allergies to study drug(s) 7. Concomitant participation in other study protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15
Dates: Start 2007-10; Study Completion 2008-07

PRIMARY OUTCOMES:
Measurement of the effect of a preemptive peripheral nerve block on the hyperalgesic response to an artificially induced sunburn.

SECONDARY OUTCOMES:
Measurement of the effect of a preemptive peripheral nerve block on the release of pro-inflammatory cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Martin S Angst, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States